CLINICAL TRIAL: NCT07060170
Title: The Effect of Augmented Reality Versus Virtual Reality Glasses as Distraction Techniques in Children During the Administration of Local Anesthesia A Randomized Clinical Trial
Brief Title: Comparing Augmented Reality and Virtual Reality Glasses to Help Children Feel Less Pain and Anxiety During Local Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riham Abbas (Other)
Responsible Party: Sponsor-Investigator, Riham Abbas, General practitioner, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: FDASU-Rec IM012411
Record Dates: First submitted 2025-02-24; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-12

CONDITIONS: Dental Anxiety; Dental Fear; Dental Fear and Anxiety
Keywords: salivary alpha amylase; dental anxiety; cortisol; Virtual Reality; Local Anesthesia; child; Behavior
MeSH Terms: conditions — Anxiety Disorders; Behavior

STUDY DESIGN:
Intervention Model Description: Teeth in each patient will be randomly assigned to receive both interventions sequentially, using a simple randomization technique. Each time a new patient is to be enrolled in the study, he\she will be asked to select a sequentially numbered sealed opaque envelop that determines which type of distraction method will be implemented first. In the subsequent treatment visit, the other distraction technique will be automatically applied, since this is a split mouth designed study.
  A set of 40 envelopes (20 envelopes for augmented reality glasses and 20 envelops for virtual reality glasses) will be kept with a third party (the main supervisor), who will not be involved in the data collection, to ensure allocation concealment.
Who Masked: Outcomes Assessor
Masking Description: The main supervisor will code the patients' tooth allocation in order to blind the statistician and the clinical pathologist who will assess the salivary biomarker levels in the samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maxillary right primary molars (Active Comparator): In this Split-mouth Randomized Controlled Trial, 5-8-year-old female and male children will be enrolled. They will receive local anesthesia on the right side of the arch using one of the distraction methods, then after one to two weeks they will receive local anesthesia on other side of the arch using a different distraction method
  Interventions: Device: Augmented Reality Glasses; Device: Virtual Reality Glasses
- Maxillary left primary molars (Active Comparator): In this Split-mouth Randomized Controlled Trial, 5-8-year-old female and male children will be enrolled. They will receive local anesthesia on the left side of the arch using one of the distraction methods, then after one to two weeks they will receive local anesthesia on other side of the arch using a different distraction method
  Interventions: Device: Augmented Reality Glasses; Device: Virtual Reality Glasses

INTERVENTIONS:
Device: Augmented Reality Glasses — The child will wear the augmented reality glass, and a cartoon movie will be displayed during the injection of local anesthesia
Device: Virtual Reality Glasses — The child will wear the glass, and a cartoon movie will be displayed during the injection of local anesthesia.

SUMMARY:
The goal of this clinical trial is to learn if audio-visual method of distraction is useful to control the pain and fear associated with dental treatment in children. The main questions it aims to answer are:

• How their body reacts-such as changes in heart rate, oxygen levels, and certain chemicals in their saliva-before and after getting local anesthesia? Researchers will test two types of glasses that display cartoons to help children feel less anxious.

Participants will:

* Have an introductory visit to be more familiar with dental environment and their cooperation will be tested.
* In the next 2 visits they will wear either of the glasses while receiving local anesthesia
* Saliva will be collected, and their heart rate and oxygen levels will be calculated each time

ELIGIBILITY:
Inclusion Criteria:

1. 5-8 year-old female and male patients.
2. Cooperative patients (rating 3 or 4 on the Frankl's Behavior Rating Scale).
3. American Society of Anesthesiologists (ASA) Class (I).
4. Patients need dental treatment under local anesthetic infiltration.
5. Patients without known anxiety disorders.
6. Patients with body weight that is considered normal according to their age and gender (95th percentile growth curve).
7. Patients without a prior history of receiving local anesthetic.
8. Patients with at least one vital primary molar with deep carious lesion on each side of the dental arch, who require to be treated under local anesthesia

Exclusion Criteria

1. Patients with special health care needs.
2. Patients on corticosteroid medications.
3. Patients having known salivary disorders, such as Sjogren's syndrome.
4. Parents who refused to sign the informed consent.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain perception and anxiety before and after local anesthesia administration using augmented reality glasses in 5-8-year-old children | Pain perception will be assessed immediately before, and immediately after local anesthetics administration.
  The Wong-Baker FACES Pain Rating Scale Arabic Version, will be used to subjectively assess the pain perception before and after local anesthetics administration, the scale uses cartoon faces representing pain levels from 0 ("no pain") to 10 ("worst pain imaginable").
Evaluation of pain perception and anxiety before and after local anesthesia administration using augmented reality glasses in 5-8-year-old children | Pain perception will be assessed from needle insertion to completion of injection (1 minute) of local anesthesia.
  The face, legs, activity, cry, consolability (FLACC) behavioral pain assessment scale will be used to objectively assess the pain perception during local anesthetics administration, this scale consists of 5 categories, each category is scored from 0 to 2, with a total score ranging from 0 ("relaxed and comfortable") to 10 ("sever discomfort or pain or both").

SECONDARY OUTCOMES:
Changes in the levels of the salivary cortisol, of 5-8-year-old children before and after the administration of local anesthesia using augmented reality glasses as a distraction | Salivary stress biomarker will be assessed at baseline, and 20 minutes after local anesthetics administration while the child is distracted using either augmented reality glasses or virtual reality glasses.
  Salivary stress biomarker (salivary cortisol) will be assessed using enzyme linked immunoassay (ELISA) technique.
Changes in the levels of the salivary alpha amylase, of 5-8-year-old children before and after the administration of local anesthesia using augmented reality glasses as a distraction | Salivary stress biomarker will be assessed at baseline, and 20 minutes after local anesthetics administration while the child is distracted using either augmented reality glasses or virtual reality glasses.
  Salivary stress biomarker (salivary alpha amylase) will be assessed using enzyme linked immunoassay (ELISA) technique.
Changes in the heart rate of 5-8-year-old children before, during, and after the administration of local anesthesia using either augmented or virtual reality glasses as a distraction | Heart rate and oxygen saturation will be assessed at baseline, at the onset anesthesia administrating, and one minute after local anesthetics administration while the child is distracted using either augmented reality glasses or virtual reality glasses
  The physiological measures of heart rate will be used to evaluate the anxiety using pulse oximeter.
Changes in the oxygen saturation of 5-8-year-old children before, during, and after the administration of local anesthesia using either augmented or virtual reality glasses as a distraction | Oxygen saturation will be assessed at baseline, at the onset anesthesia administrating, and one minute after local anesthetics administration while the child is distracted using either augmented reality glasses or virtual reality glasses
  The physiological measures of oxygen saturation will be used to evaluate the anxiety using pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Professor of Pediatric Dentistry and Dental Public Health, Study Director — Faculty of Dentistry, Ain Shams University; Lecturer of Pediatric Dentistry and Dental Public Health, Study Director — Faculty of Dentistry, Ain Shams University
Locations (1):
- Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Ain Shams University, Cairo, Egypt, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No
Faculty of Dentistry Ain Shams University Research Ethics Committee, state that data will not be shared to preserve the confidentiality.

REFERENCES:
- [Background] Singh Y, Parameshwarappa P, Mathew MG, Meghana SB, Kenchappa M, Nagaveni NB. Comparison of distraction techniques using salivary biomarkers during local anaesthesia administration in children aged 3-5 years: A clinical study. Indian J Dent Res. 2023 Apr-Jun;34(2):169-173. doi: 10.4103/ijdr.ijdr_132_22. PMID 37787206
- [Background] Subramaniam SD, Doss B, Chanderasekar LD, Madhavan A, Rosary AM. Scope of physiological and behavioural pain assessment techniques in children - a review. Healthc Technol Lett. 2018 Jul 17;5(4):124-129. doi: 10.1049/htl.2017.0108. eCollection 2018 Aug. PMID 30155264
- [Background] Sharma Y, Bhatia HP, Sood S, Sharma N, Singh A. Effectiveness of Virtual Reality Glasses Digital Screens and Verbal Command as a Method to Distract Young Patients during Administration of Local Anesthesia. Int J Clin Pediatr Dent. 2021;14(Suppl 2):S143-S147. doi: 10.5005/jp-journals-10005-2094. PMID 35645477
- [Background] Rao DG, Havale R, Nagaraj M, Karobari NM, Latha AM, Tharay N, Shrutha SP. Assessment of Efficacy of Virtual Reality Distraction in Reducing Pain Perception and Anxiety in Children Aged 6-10 Years: A Behavioral Interventional Study. Int J Clin Pediatr Dent. 2019 Nov-Dec;12(6):510-513. doi: 10.5005/jp-journals-10005-1694. PMID 32440065
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857